CLINICAL TRIAL: NCT06296303
Title: Effect of Pulsed Magnetic Therapy Versus Phonophoresis on Sciatic Nerve Cross Section Measured by Ultrasonography in Discogenic Lumbar Radiculopathy Patients
Brief Title: Effect of Pulsed Magnetic Therapy Versus Phonophoresis in Discogenic Lumbar Radiculopathy Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Badr Hassanein, MSc, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MBH24
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Lumbar Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pulsed electromagnetic therapy group (Experimental): Patients in this group will receive Pulsed electromagnetic therapy + Conventional physical therapy
  Interventions: Other: Pulsed electromagnetic therapy; Other: Conventional physical therapy
- Ultrasound phonophoresis group (Experimental): Patients in this group will receive Ultrasound phonophoresis + Conventional physical therapy
  Interventions: Other: Ultrasound phonophoresis; Other: Conventional physical therapy
- Control group (Active Comparator): Patients in this group will receive Conventional physical therapy
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Pulsed electromagnetic therapy — Pulsed etromagnetic therapy (1000 gauss) on sciatic nerve in gluteal fold. ( 30 min )
  Arms: Pulsed electromagnetic therapy group
Other: Ultrasound phonophoresis — Phonophoresis using dexamethasone and topical diclofenac sodium gel on sciatic nerve in subgluteal fold and mid thigh
  Arms: Ultrasound phonophoresis group
Other: Conventional physical therapy — Conventional physical therapy consisting of
  1. IF current on lumbar spine. (15 min )
  2. Hotpack on lumbar spine . (15 min )
  3. Neurodynamic mobilization .
  4. Mobilization and manipulation for lumbar spine.
  5. Exercises

SUMMARY:
Purposes of the study

To investigate the effect of pulsed magnetic therapy versus phonophoresis in discogenic lumbar radiculopathy patients

DETAILED DESCRIPTION:
Patients will be randomized into either pulsed magnetic therapy group or phonophoresis group. Patients will receive the intervention for six weeks. Outcomes will be assessed at baseline and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ranges from 20 -45
* Unilateral chronic lumbosacral radiculopathy
* Intervertebral disc herniation confirmed by MRI
* one of the following :

  1. H- reflex amplitude side to side difference 0.67 in absence of latency difference.
  2. H- reflex amplitude side to side difference smaller than 0.5 in p of latency difference.

  3 - Side to side H- reflex latency difference more than 1 msec. 4- Prolonged H-reflex latency more than 30 msec.

Exclusion Criteria:

* Systematic disease
* Lumbar canal stenosis
* Pervious surgeries
* Scoliosis
* Kyphosis
* Spinal fracture
* Bilateral symptoms
* Steroid injection

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-03 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain | Change from Baseline pain and function at 6 weeks
  Visual analogue scale
Disability | Change from Baseline pain and function at 6 weeks
  Oswestry disability index
Sciatic nerve cross sectional area | Change from Baseline pain and function at 6 weeks
  Diagnostic Ultrasound

SECONDARY OUTCOMES:
H-reflex amplitude | Change from Baseline pain and function at 6 weeks
  by EMG unit
H-reflex side-to-side amplitude (H/H) ratio | Change from Baseline pain and function at 6 weeks
  by EMG unit

IPD SHARING:
Plan to Share IPD: Undecided